CLINICAL TRIAL: NCT02873065
Title: Efficacy and Safety of 1-week Triple Therapy With Ilaprazole for the Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LivzonIY-81149R-11-02
Record Dates: First submitted 2016-07-26; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Helicobacter Pylori Eradication
MeSH Terms: interventions — ilaprazole; Amoxicillin; BID protein, human; Clarithromycin

ARMS (2):
- Ilaprazole (Experimental): Ilaprazole -based quadruple therapy for 7days：Ilaprazole -based quadruple therapy for 7days: Ilaprazole 5mg bid.
  Interventions: Drug: Ilaprazole
- Esoprazole (Active Comparator): Esoprazole -based quadruple therapy for 14 days: Esoprazole 20mg bid.
  Interventions: Drug: Esoprazole

INTERVENTIONS:
Drug: Ilaprazole
  Other Names: Ilaprazole and amoxicillin 1000mg bid, clarithromycin 500mg bid
  Arms: Ilaprazole
Drug: Esoprazole
  Other Names: Esoprazole and Bismuth Potassium Citrate 220mg bid, Amoxicillin 1000mg bid, Clarithromycin 500mg bid
  Arms: Esoprazole

SUMMARY:
This study compared efficacy and safety of Ilaprazole based triple regimen therapy including Ilaprazole 5mg, Clarithromycin 500mg and Amoxicillin Cap(Amoxicillin) 1000mg BID on the first line eradication treatment of H.pylori

DETAILED DESCRIPTION:
Participants are defined as persons who have endoscopically confirmed on gastric or duodenal ulcer(including scar stage) ,gastritis and dyspepsia confirmed to be H.pylori positive patients in the biopsy and UBT test. For 7 days, Participants treated as Esoprazole based triple regimen therapy therapy including Esoprazole 20mg，Clarithromycin 500mg and Amoxicillin Cap(Amoxicillin) 1000mg BID. After treatment, The healing rate was evaluated in the UBT test and Biopsy at 49±5days from the first day dosing

ELIGIBILITY:
Inclusion Criteria:

* Subject must have endoscopically confirmed on gastric, duodenal ulcer(including scar) or gastritis confirmed to be H.pylori positive patients in the biopsy and UBT test.
* Subject who fully understands conditions of clinical trial.
* Subject who agrees to participate and spontaneously sign the ICF

Exclusion Criteria:

* Known hypersensitivity to any component of ilaprazole, Esoprazole, Amoxicillin and Clarithromycin
* Subjects who are taking contraindicated medications for experimental and concomitant drug
* Administrated of PPI, antibiotic medication within 4 weeks prior to commencement of the study
* Pregnant and/or lactating women
* Reproductive aged women not using contraception
* Uncontrolled diabetics
* Uncontrolled hypertension
* Uncontrolled liver dysfunction
* Alcoholics
* Subjects with a history of digestive malignancy within 5 years
* Subjects with a history of gastrectomy or esophagectomy
* Subjects with hereditary diseases such as Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption
* Subjects participating in a clinical trial before another trial within 30 days
* Inconsistent judged subject by researcher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori as assessed by UBT test | 4 weeks

SECONDARY OUTCOMES:
Frequency of side effects of each treatment | 2 months